CLINICAL TRIAL: NCT00795444
Title: Pilot Study Of The Effect Of A CCR5 Coreceptor Antagonist On The Latency And Reservoir Of HIV-1 In Patients Taking Highly Active Antiretroviral Therapy
Brief Title: Effect Of A CCR5 Coreceptor Antagonist On The Latency And Reservoir Of HIV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERRADVIH-01; Eudra CT 2007-003995-21
Record Dates: First submitted 2008-11-10; First posted 2008-11-21 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: HIV-1
Keywords: HIV-1; CCR5 coreceptor antagonist (Maraviroc); the cell reservoir of HIV-1
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc (Experimental): Adult patients with HIV infection and a viral load that has been suppressed for a long period (less than 50 copies/mL for at least 2 years) while on antiretroviral therapy.The treatment group will maintain the habitual antiretroviral therapy combined with maraviroc.
  Interventions: Drug: maraviroc

INTERVENTIONS:
Drug: maraviroc — Maraviroc (INN), 300 mg tablets. A dose of 300 mg will be administered every 12 hours.
  Other Names: celsentri; CCR5 coreceptor antagonist

SUMMARY:
The presence of a pool of cells latently infected by HIV-1 in patients taking HAART and with a viral load below 50 copies/mL is the main limitation to eradication of the virus from the body. This viral reservoir prevents antiretroviral therapy from being interrupted; therefore, patients are obliged to continue with treatment for a period calculated to be greater than 60 years.

Despite the important advances in knowledge of the biology of this reservoir, we still have no real knowledge about its dynamics. The opportunity to carry out a clinical trial for the first time with CCR5 coreceptor antagonists is exceptional, since the results could provide important information on the nature of this reservoir.

If maintenance of the reservoir is a dynamic process, inclusion of CCR5 inhibitors is expected to lead to a reduction in the size of this reservoir. This effect could be critical when including IAT (viral reactivation), since, in theory, it would be necessary to act on a smaller reservoir. Current consensus is that it would be necessary to act on almost 100% of the viral reservoir (approximately 1,000,000 cells).

The study has also been designed to enable us to understand the biochemical and molecular mechanisms by which certain drugs can induce viral reactivation in vitro as a previous step to a clinical trial aimed at reactivating viral latency and eradicating HIV-1 from the body.

ELIGIBILITY:
Inclusion Criteria:

* After receiving information on the design and objectives of the study, the possible risks involved, and the fact that they can refuse to collaborate at any time, patients will give their informed consent to participate in the study and agree to provide material for the cellular and molecular studies.
* Aged over 18 years.
* Chronic HIV infection
* Antiretroviral therapy with at least 3 drugs for at least 2 years and with no modifications expected during the study. Antiretroviral drugs can be switched due to intolerance as long as plasma viremia remains controlled.
* Undetectable viral load determined by ultrasensitive techniques (<50 copies HIV RNA/mL) for at least 2 years.
* CD4+ T lymphocyte count above 350 cells/mm3.
* Demonstration of R5 viral tropism (use of CCR5 coreceptors) by phenotyping in plasma samples stored before antiretroviral therapy is started.
* Understand the objective of the study and be available to make frequent visits to the hospital.

Exclusion Criteria:

* Previous failure of antiretroviral therapy, understood as a rebound in viral load that can be detected after having reached undetectable levels. Low-grade increases (<200 copies of HIV RNA/mL) and transitory increases (blips) resolved without modifying antiretroviral therapy are excluded.
* Proven resistance against the antiretroviral drugs under study.
* Planned interruption of antiretroviral therapy.
* Taking immunosuppressive or immunostimulating medication of any type, including valproic acid.
* Taking a fusion inhibitor (enfuvirtide).
* Pregnancy or intention to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Frequency of resting CD4+ T cells infected by a replicative virus | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno Guillen, MD,PhD, Principal Investigator — HOSPITAL UNIVERSITARIO RAMON Y CAJAL. MADRID
Locations (1):
- Hospital Universitario Ramon Y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Serrano-Villar S, Gutierrez C, Vallejo A, Hernandez-Novoa B, Diaz L, Abad Fernandez M, Madrid N, Dronda F, Zamora J, Munoz-Fernandez MA, Moreno S. The CD4/CD8 ratio in HIV-infected subjects is independently associated with T-cell activation despite long-term viral suppression. J Infect. 2013 Jan;66(1):57-66. doi: 10.1016/j.jinf.2012.09.013. Epub 2012 Oct 6. PMID 23046968
- [Derived] Gutierrez C, Diaz L, Vallejo A, Hernandez-Novoa B, Abad M, Madrid N, Dahl V, Rubio R, Moreno AM, Dronda F, Casado JL, Navas E, Perez-Elias MJ, Zamora J, Palmer S, Munoz E, Munoz-Fernandez MA, Moreno S. Intensification of antiretroviral therapy with a CCR5 antagonist in patients with chronic HIV-1 infection: effect on T cells latently infected. PLoS One. 2011;6(12):e27864. doi: 10.1371/journal.pone.0027864. Epub 2011 Dec 8. PMID 22174752